CLINICAL TRIAL: NCT04885062
Title: Belun Ring Platform (BLS-100) Home Sleep Apnea Testing Device With an Improved Algorithm for Assessment of Obstructive Sleep Apnea: A Comparison to In-Lab Polysomnography
Brief Title: Belun Ring Platform With an Improved Algorithm for OSA Assessment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Belun Technology Company Limited (Other)
Collaborators: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY20201259
Record Dates: First submitted 2021-05-04; First posted 2021-05-13 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Sleep-Disordered Breathing; Sleep Architecture
Keywords: Obstructive Sleep Apnea; Wearable; Home Sleep Apnea Testing; Photoplethysmography; Validation; Artificial Intelligence
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- UH-Participant (Experimental): Potential participants with suspected OSA will be identified from the schedule of the UH Beachwood and Bolwell sleep labs.Those subjects who satisfy the study inclusion and exclusion criteria will be approached and invited to participate in the study.
  Interventions: Device: Belun Ring; Diagnostic Test: PSG

INTERVENTIONS:
Device: Belun Ring — The Belun Ring sensor will be applied to the proximal phalanx of the index finger in the non-dominant hand of the participating individuals prior to their sleep onset in the sleep lab and will be removed upon awakening at the end of the sleep period on the following morning. The attended in-lab sleep study will be performed simultaneously in a standard fashion.
Diagnostic Test: PSG — All patients scheduled for attended overnight in-lab polysomnography (PSG) in our 2 sleep labs will undergo PSG testing. On the same night of the PSG testing, these same patients will also wear the Belun Ring device. After the study, we will compare results of the Belun Ring device vis-à-vis with the results of the PSG on the same patient.

SUMMARY:
OSA is commonly diagnosed with either attended in-lab polysomnography (PSG) or unattended home sleep apnea testing (HSAT). The BLS-100 (Belun Technology Company Limited, Hong Kong) is a novel neural network-based HSAT platform consists of a ring shape pulse oximeter sensor, a cradle, and an improved proprietary analytic algorithm. This study investigates the hypothesis that the BLS-100 is a reasonable HSAT device for OSA assessment.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form.
* Age 18-80
* Clinically assessed and suspicious for OSA

Exclusion Criteria:

* Full night PAP titration study
* On home O2, noninvasive ventilator, diaphragmatic pacing, or any form of nerve stimulator
* Having atrial fibrillation-flutter, pacemaker/defibrillator, LVEF < 55%, left ventricular assist device (LVAD), or status post cardiac transplantation
* Patients taking narcotics
* Recent hospitalization or recent surgery in the past 30 days
* Unstable cardiopulmonary status on the night of the study judged to be unsafe for sleep study by the sleep tech and/or the on-call sleep physician

An individual who meets the above criteria but fails to have at least 4 hours of technically valid sleep based on BLS-100 in a diagnostic study or at least 3 hours of technically valid sleep during the diagnostic portion of a split night study will be excluded from statistical analyses.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
REI parameters | 1 year
  To determine the overall accuracy, sensitivity, and specificity of the BLS-100 in assessing OSA by comparing to the attended in-lab PSG in individuals referred to the sleep labs with clinical suspicion of OSA.

SECONDARY OUTCOMES:
Sleep stage parameters | 1 year
  To determine the accuracy of BLS-100 sleep stage parameters to classify the human sleep stage (Wake, REM and Non-REM) by comparing to the classification results of in-lab PSG.

CONTACTS AND LOCATIONS:
Overall Officials: Ambrose A Chiang, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No